CLINICAL TRIAL: NCT05880329
Title: Feasibility Cohort Study on Predictors of Diagnosis and Prognosis of Urine Infection in Care Home Residents: DIagnoSing Care hOme UTI Study
Brief Title: DIagnoSing Care hOme UTI Study
Acronym: DISCO UTI
Status: Recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: University of Oxford (Other); University of Bristol (Other); Public Health Wales (Other Government)
Responsible Party: Sponsor
Other Study IDs: 79003
Record Dates: First submitted 2023-03-07; First posted 2023-05-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples.
  We intend to seek further funding to complete pilot sequencing work on the urine microbiome from some of the samples collected, including any carriage of antimicrobial resistance genes. After use in DISCO UTI, samples would be spun and frozen, then couriered and stored at the University of Oxford.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Care home residents: 100 care home residents will be recruited and followed up for 6 months.
  Interventions: Diagnostic Test: Candidate POCTs for detecting UTI

INTERVENTIONS:
Diagnostic Test: Candidate POCTs for detecting UTI — POCT performance will be evaluated in participants who experience possible UTI.

SUMMARY:
The number of care home residents is increasing and urinary tract infections (UTIs) are common amongst this group. Accurate diagnosis of UTI is important because not treating an infection may lead to serious consequences including death. However, giving antibiotic treatment when there isn't an infection causes side effects and antibiotic resistance, making future infections harder to treat.

Unfortunately, there are several challenges that mean that it is difficult to diagnose UTI accurately in care home residents. Firstly, UTIs don't always cause clear symptoms for people who live in care homes. They sometimes just cause symptoms like confusion which can have lots of different possible causes. Secondly, it may be hard for people living with dementia to say how they are feeling or to easily provide a urine sample. Thirdly, many people who live in care homes have bacteria present in their urine even when they are well, but this not harmful and does not need treatment. Finally, urine tests that are currently available do not give accurate or quick results.

We have thought about some new ways that might help show us if someone in a care home really has a UTI but we don't know yet whether these will work. Our ideas include 1) Working out which symptoms or signs mean a UTI is more likely 2) Detecting new markers of infection in urine samples and 3) Trying out new bedside tests that give rapid results.

For this study we plan to recruit 100 care home residents who will be followed up over 6 months. All 100 participants will provide information and a urine sample at the beginning of the study. 25 of these participants will also provide repeated weekly samples for 4 weeks to look at any changes in the urine over time. Additional information and urine samples will be collected if a participant develops a possible UTI during the study and any treatments will be recorded.

Our findings will be used to develop a funding application for a larger study aiming to improve the diagnosis of UTI in care home residents.

DETAILED DESCRIPTION:
This feasibility observational study will be conducted in four overlapping stages: recruiting a cohort of 100 care home residents (CHR) from up to 10 care homes across the Thames Valley and Wessex (Stage 1); collecting weekly repeated baseline urine samples from a subset of participants (without suspected UTI) (Stage 2); following all 100 participants for 6 months and collecting additional data on those who develop possible UTI (Stage 3), and interviewing participants, their families and care home staff about study feasibility and acceptability (Stage 4).

Stage 1 - Cohort recruitment and baseline data collection

Baseline assessments:

Following consent, baseline data will be collected including demographics, medical history, and a description of baseline functional ability. We will also collect a urine sample for baseline microbiological and urinary biomarker analyses for each participant.

Stage 2 - Repeat urine sampling cohort 25 CHR recruited in Stage 1 will be asked to provide weekly urine samples for four weeks. Urine samples will be sent for microbiological and urinary biomarker analyses.

CHR who develop a possible UTI during this stage will contribute to Stage 3 and will continue to have any remaining weekly samples collected if possible.

Stage 3 - Possible UTI episodes All 100 CHR recruited during Stage 1 will be followed for 6 months. Care home staff will be asked to alert the research team as soon as any participant in the cohort develops possible UTI. This would include any situation where care home staff have decided to consult with a healthcare professional because they have detected a change in the CHR or their urine and believe that a UTI is 'a likely cause'. This would not include residents who become acutely unwell from a source that is clearly not UTI at onset (e.g. chest or skin infection or cerebrovascular event).

Participants who experience possible UTI will have a 'symptomatic baseline' assessment and follow up visits at 14 and 28 days. A urine sample will be collected. If possible and this doesn't delay care, this will be before any treatment is initiated. Repeat urine samples will be collected at days 14 and 28.

Some of the urine taken at symptomatic baseline and day 28 will also be tested using one or more novel POCTs by a member of the research team.

Stage 4 - Qualitative sub-study We will conduct a qualitative evaluation to explore study acceptability and barriers and facilitators to study procedures. Care home staff, residents, and their families will be asked to participate in semi-structured interviews towards the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for the study, or if lacking capacity, a consultee willing to complete a consultee declaration form.
* Permanently living in a care home (nursing, residential or mixed).
* Aged 65 or over.

Exclusion Criteria:

* Current/recent suspected UTI (within last 4 weeks). However, may be reassessed for eligibility after 4 weeks.
* Temporary/respite resident (unlikely to remain living in the care home for the 6 months of the study duration)
* Terminal illness limiting life expectancy such that inclusion would be inappropriate (as judged by care home staff).
* Known to have a medical condition or be on treatment that is likely to result in severe impairment of the immune system. For example, neutropenia, recent cancer chemotherapy or radiotherapy, or long-term use of oral steroids or other immunosuppressant medication.
* Experiencing faecal incontinence to the extent that it is impossible to obtain an uncontaminated urine sample (as determined by care home staff).
* Indwelling urinary catheter or regular use of intermittent catheterisation.
* Structural urological abnormalities. For example, renal polycystic disease, horseshoe kidney, hydronephrosis, renal hypoplasia
* Current renal tract malignancy. However, residents with prostate cancer will be eligible if they do not require catheterisation and are not considered terminally ill.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: We aim to recruit a cohort of 100 care home residents over 65 years of age from up to 10 care home sites.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
As a feasibility study, there is no primary outcome measure. | Baseline

SECONDARY OUTCOMES:
Proportion of care homes agreeing to participate when recruiting care homes as research sites. | Baseline
Proportion of residents screened that are eligible and proportion of eligible that are recruited. | Baseline
Proportion of baseline urine samples obtained from participants recruited (consented) | Baseline
Proportion of repeated urine samples obtained of those participating in Stage 2 | 2, 3 and 4 weeks
Quality of urine samples obtained | Through study completion, 6 months
  Proportions of samples collected mid-stream clean catch, vs other collection techniques Proportions of samples contaminated (as reported by staff collecting samples) Proportions of samples with microbiological evidence of contamination
Adherence to urine transport protocols | Through study completion, 6 months
  Time from sampling until receipt in laboratory Proportion recorded as stored refrigerated prior to transportation
Proportion of residents that experience a possible UTI during the follow-up period that are reported to the research team. | Through study completion, 6 months
Proportion of residents with possible UTI that are not reported to the research team. | Assessed weekly through to study completion at 6 months
Proportion of residents with possible UTI in whom the following is obtained: | Through study completion, 6 months
  * Symptomatic baseline data on the characteristics of the possible UTI
  * A urine sample at onset of possible UTI
  * A urine sample prior to any antibiotic administration
  * Follow-up data
  * Follow-up urine samples at 14 and 28 days from symptom onset
Using semi-structured interviews with qualitative analysis to describe the views of care home staff, participants and family members on: | Through study completion, 6 months
  1. Barriers and facilitators to taking part in the study.
  2. Experience of obtaining/giving consent.
  3. Experience of being a participant/family member of a participant.
  4. Experience of giving/collecting urine samples including resident and staff willingness and capacity to obtain weekly urine samples.
  5. Experience of reporting a possible UTI to the study team and any barriers or facilitators to reporting in a timely fashion.
  6. The diagnosis of UTI and how this is determined in usual care
  7. The diagnosis of UTI and how this was determined during the study
  8. Additional tests including POCTs for UTI
Participant baseline demographic characteristics predictive of subsequent possible UTI/clinical outcomes | Through study completion, 6 months
Participant clinical characteristics at point of possible UTI and association with clinical outcomes | Through study completion, 6 months
Changes in weekly sample microbiology | Baseline, 2, 3 and 4 weeks
  Description of any changes in the microbiological results of samples sent weekly from weeks 1-4
Predictors of weekly sample microbiology and changes in microbiology | Baseline, 2, 3 and 4 weeks
  Including previous urine culture results, resident demographic characteristics, and sampling characteristics
Association between asymptomatic bacteriuria at baseline or in weekly sampling and onset of possible UTI during follow up period | Through study completion, 6 months
Association of each urinary biomarker with asymptomatic bacteriuria | Baseline
  Assess whether concentration of biomarkers listed below is associated with asymptomatic bacteriuria:
  Matrix metallopeptidase-9, neutrophil gelatinase associated lipocalin (NGAL), Interleukin , Interleukin 8, Interleukin 6, Interleukin 6, Interleukin 10, secretory IgA, and chemokine (C-X-C motif) ligand 1
Urinary biomarker concentrations in urine samples from asymptomatic participants without bacteriuria | Baseline
  Matrix metallopeptidase-9, neutrophil gelatinase associated lipocalin (NGAL), Interleukin , Interleukin 8, Interleukin 6, Interleukin 6, Interleukin 10, secretory IgA, and chemokine (C-X-C motif) ligand 1
Urinary biomarker concentrations in urine samples from possible UTI episodes | Through study completion, 6 months
  Matrix metallopeptidase-9, neutrophil gelatinase associated lipocalin (NGAL), Interleukin , Interleukin 8, Interleukin 6, Interleukin 6, Interleukin 10, secretory IgA, and chemokine (C-X-C motif) ligand 1
Failure rate of the POCT in residents with possible UTI (no result or invalid result) | Through study completion, 6 months
Agreement between POCT result and laboratory enhanced culture result at symptom onset for each possible UTI episode, and at 28 days post symptom on set | Through study completion, 6 months
  Comparison to be made between each POCT result and the result from the enhanced culture carried out in the laboratory at symptomatic baseline and 28 day follow up of each possible UTI episode.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Moore, Principal Investigator — University of Oxford; Nick Francis, Principal Investigator — University of Oxford
Locations (1):
- Solent NHS Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this stage.